CLINICAL TRIAL: NCT01092455
Title: Citrasate® Effect On Heparin N Requirements During Hemodialysis Treatment: A Phase IV,Study to Investigate the Effects of Citrasate on Heparin N Requirements During Hemodialysis Treatment in Subjects Maintained on Thrice Weekly Hemodialysis
Brief Title: Multi-center Study to Investigate the Effects of Citrasate® on Heparin N Requirements During Hemodialysis Treatment
Status: Completed | Type: Observational
Sponsor: Randolph Quinn (Industry)
Responsible Party: Sponsor-Investigator, Randolph Quinn, Manager, Regulatory Affairs, Fresenius Medical Care North America
Organization: Fresenius Medical Care North America (Industry)
Other Study IDs: 208-09
Record Dates: First submitted 2010-03-11; First posted 2010-03-25 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Renal Dialysis
Keywords: End Stage Renal Disease; Renal Dialysis; Hemodialysis therapy; Heparin; Citrasate; Anticoagulant
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Citrasate and heparin reduction: Sequential hemodialysis treatment study in which all enrollees move through four (4) separate treatment phases. Results from the separate phases will be compared to standard bicarbonate dialysis with standard does of heparin.
  Interventions: Drug: Heparin N reduction

INTERVENTIONS:
Drug: Heparin N reduction — Dialysis with Citrasate, acid concentrate plus 100% of patient's standard heparin N dose; Dialysis with Citrasate acid concentrate plus 80% of patient's standard heparin N dose; Dialysis with Citrasate acid concentrate plus 66.7% of patient's standard heparin N dose.
  Other Names: Citrasate®; Heparin N

SUMMARY:
The purpose of this study is to determine whether the use of Citrasate®, citric acid dialysate enables the reduction of the heparin N (anticoagulant) dose in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
During hemodialysis, waste products are removed from the blood by diffusion across the dialyzer membrane into an electrolyte solution known as dialysate. Dialysate is produced from acid concentrate, bicarbonate solution and water using a three stream proportioning system that mixes the acid concentrate, bicarbonate and water to produce the final dialysate. Patients are typically anticoagulated with heparin during dialysis to prevent blood from clotting in the extracorpoeial circuit. Heparin use is associated with significant risks including the possibility of bleeding, heparin induced thrombocytopenia (HIT) and contamination. For these reasons, the possibility of reducing heparin dose while maintaining HD adequacy is clinically attractive. Citrasate® is an FDA approved acid concentrate that contains citric acid (citrate) rather than acetic acid (acetate) which is traditionally used in acid concentrate. Citrate in higher concentrations is also a known anticoagulant. We are therefore conducting this study to determine whether the use of Citrasate, citric acid dialysate enables the reduction of the heparin requirements in patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is capable of giving informed consent, or has an acceptable surrogate capable of giving consent on the subject's behalf.
* ESRD maintained on thrice weekly HD
* Stable Heparin prescription (Heparin dose) for the previous 4 weeks
* Dialyzed using bolus heparin anticoagulation with dose >/= 2000 units per treatment
* Hgb >/= 9.5 prior to study start
* eKt/V >/= 1.0 (or spKt/V >/= 1.2) in the monthly lab work prior to study start

Exclusion Criteria:

* Any laboratory abnormality, medical condition or psychiatric disorder which in the opinion of the investigator would put the subject's disease management at risk or may result in the subject being unable to comply with study requirements
* Patient is maintained on Coumadin therapy or LMW heparin
* Known history of HIT, coagulopathy or any other bleeding and/or thrombotic disorders
* Patients dialyzed with < 2000 units of Heparin per treatment
* Dialyzed without heparin
* Known pregnancy
* Dialyzed with reuse of hemodialyzers
* Documented clotted dialyzer or dialysis lines in last 30 days (1 month) requiring changing dialyzer, bloodlines or terminating treatment
* Randomized in a clinical trial involving anticoagulation in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the hemodialysis population in the participating facilities (study sites).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of dialyzer conductivity clearance (KECN) when dialyzed with Citrasate, acid concentrate and 80% of baseline Heparin dose compared to dialysis using standard bicarbonate dialysate and standard dose heparin N (baseline). | Baseline and 6 months

SECONDARY OUTCOMES:
Non-inferiority of conductivity clearance when dialyzed with Citrasate and 66.7% baseline Heparin dose as compared to baseline. | Baseline and 6 months
Dialyzer or system clotting with Citrasate plus reduced Heparin compared to baseline. | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Sands, MD MMM, Study Director — Fresenius Medical Care North America
Locations (8):
- United States (8):
  - Avantus Renal Therapy-Saint Raphael Dialysis Center, New Haven, Connecticut
  - Irving Place Dialysis Center, New York, New York
  - Upper Manhattan Dialysis Clinic, New York, New York
  - Yorkville Dialysis Center, New York, New York
  - DaVita Medical Center Houston, Houston, Texas
  - DaVita Rivercenter Dialysis Clinic, San Antonio, Texas
  - DaVita Downtown Dialysis Clinic, San Antonio, Texas
  - DaVita Northwest Medical Center, San Antonio, Texas